CLINICAL TRIAL: NCT05498519
Title: A Phase I, Open-Label, Multi-Center, Dose-escalation/ Dose-expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Anti-Tumor Activity of SY-4798 Tablet in Patients With Advanced Solid Tumor
Brief Title: A First-in-Human, Phase 1 Study of SY-4798 in Patients With Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shouyao Holdings (Beijing) Co. LTD (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SY-4798-I-01
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Advanced Solid Tumor
Keywords: SY-4798; FGFR4; Advanced solid tumor; FGF19+ advanced tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose-escalation and Dose-expansion (Experimental): SY-4798 will be given orally in ascending doses (escalation cohort) until the DLT or RP2D is reached. In dose-expansion phase, preliminary anti-tumor activity will be assessed in FGF19+ advanced tumor.
  Interventions: Drug: SY-4798

INTERVENTIONS:
Drug: SY-4798 — FGFR4 selective inhibitor
  Other Names: SY-4798 Tablet

SUMMARY:
This is a Phase 1, open-label and multicenter study of SY-4798, a highly specific and potent inhibitor of FGFR4, in patients with advanced solid tumor. This study has two phases: dose-escalation phase and dose-expansion phase.

DETAILED DESCRIPTION:
Dose-escalation phase is designed to determine the DLTs (Dose-limiting toxicity) and recommended phase II dose (RP2D) and characterize the safety, tolerability, pharmacokinetics (PK) and Pharmacodynamics (PD) of SY-4798. Other dose regimens may be explored based on the analysis of emerging PK and safety data. At this study phase, SY-4798 will be administered orally once daily (QD) in 28-day treatment cycles to adult patients with advanced solid tumor.

Dose-expansion phase is designed to evaluate the anti-tumor activity (ORR and DOR) of SY-4798 in patients with FGF19+ advanced tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 18 years at the time of screening.
2. Eastern Collaboration Oncology Group (ECOG) performance status (PS) scored of 0-1.
3. Escalation Part: Patients must have histological or cytological confirmed advanced solid tumor, which is refractory or inappropriate at this stage to standard therapies or for which no standard therapy exists. In this part, patients with hepatocellular carcinoma (HCC) and Child-Pugh scores of ≤7 are preferred.
4. Expansion Part: Patients must have histological or cytological confirmed and FGF19 IHC+ advanced solid tumor (patients with HCC should have Child-Pugh scores of ≤7), which is refractory to or inappropriate at this stage to standard therapies or for which no standard therapy exists.
5. Estimated Life expectancy ≥ 12 weeks.
6. Must have at least one assessable lesion in dose-escalation part and one measurable lesion in dose-expansion part per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1;
7. Adequate organ function as defined in the below:

   Hepatic function

   Total serum bilirubin (TBIL) ≤ 1.5 times upper limit of normal (ULN); Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 times ULN if no demonstrable liver metastases, or ≤ 5 times ULN in the presence of liver metastases/ in HCC patients.

   Bone marrow function (no blood transfusion or hematopoietic stimulator treatment within 14 days)

   Absolute neutrophil count (ANC) ≥ 1.5 x 109/L; Platelets (PLT) count ≥ 75×109/L; Hemoglobin (Hb) ≥ 85 g/L

   Renal function

   Creatinine clearance ≥ 45 mL/min.

   Coagulation function

   International standardized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN.
8. Female patients with reproductive potential must have a negative serum pregnancy test within 7 days prior to starting trial treatment, male and female patients of childbearing potential must be willing to completely abstain or agree to use an appropriate method of contraception during the entire study duration and for at least 3 months after the last dose of study medication.
9. Willingness and ability to give informed consent and follow protocol procedures, and comply with follow-up visit requirements.

Exclusion Criteria:

Patients with any of the following are excluded:

1. Patients who received chemotherapy, radiotherapy, biological therapy, endocrine therapy, immunotherapy, and other anti-tumor treatment within 4 weeks before the first administration, except for the following: Nitrosourea or mitomycin C was received within 6 weeks before the first administration; Oral fluoropyrimidines and small molecule targeted drugs within 2 weeks or 5 half-lives of the drug (whichever is longer) prior to the first administration; Chinese proprietary medicines with anti-tumor indications were received within 2 weeks before the first administration.
2. Received other unmarketed investigational drugs or treatments within 4 weeks prior to the first administration.
3. Have undergone major organ surgery (excluding needle biopsy) or had significant trauma within 4 weeks prior to the first administration.
4. Have received the treatment of FGFR4 selective or pan-FGFR inhibitors.
5. Adverse effects of previous antitumor therapy have not recovered to CTCAE 5.0 grade ≤1 (except toxicities that the investigator judged to be of no safety risk, such as alopecia, grade 2 peripheral neurotoxicity, and stable hypothyroidism with hormone replacement therapy).
6. Patients with central nervous system metastasis or meningeal metastasis with clinical symptoms, or other evidence indicates that the patient's central nervous system metastasis or meningeal metastasis has not been controlled, and those who are judged by the investigators to be unsuitable for inclusion.
7. Patients with active infection who need systematic anti-infective therapy.
8. History of immunodeficiency, including positive HIV antibody test.
9. Active hepatitis B (HBV-DNA > 103 copies/mL or 200 IU/ mL; HBV-DNA> 104 copies/mL or 2000 IU/ mL for patients with HCC), antiviral therapies except interferon are allowed. Hepatitis C virus infection (HCV-RNA >ULN).
10. A history of serious cardiovascular and cerebrovascular disease, including but not limited to: Severe cardiac rhythm and conduction abnormalities, such as ventricular arrhythmias and degree II-III atrioventricular block requiring clinical intervention; Longer QT interval at rest (QTc > 480 msec) obtained from 3 electrocardiograms (ECGs); Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or higher cardiovascular and cerebrovascular events occurred within 6 months prior to first administration; Heart failure with the New York Heart Association (NYHA) Heart function rating ≥ II or left ventricular ejection fraction (LVEF) < 50%; Clinically uncontrolled hypertension.
11. Uncontrolled effusion in the third space, not suitable for entry as determined by the investigator.
12. Patient used CYP3A4 potent inhibitors or potent inducers within 7 days before enrollment.
13. Unable to swallow or conditions that seriously affects gastrointestinal absorption as judged by the investigator.
14. Known alcohol or drug dependence.
15. Patients with mental disorders or poor compliance.
16. Pregnant and/or lactating individuals.
17. The investigator considered that the subjects had a history of other serious systemic diseases or other reasons that made them unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | Escalation Cycle 1 (28 days)
  Maximum Tolerated Dose(s) (MTD(s)) and/or recommended phase 2 dose (RP2D(s)) in Cycle 1.
Incidence of adverse events (AEs) and serious adverse events (SAEs) | Up to 24 months
  Characterization of the safety and tolerability as determined by changes in laboratory values and electrocardiograms.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) as assessed by RECIST 1.1 criteria | Up to 24 months
  Preliminary measure of anti-tumor activity of SY-4798 in patients with FGF19+ advanced tumor.
Duration of response (DOR) | Up to 24 months
  Preliminary measure of anti-tumor activity of SY-4798 in patients with FGF19+ advanced tumor.
Pharmacokinetics (Cmax) for SY-4798 | Protocol-defined time points during Cycles 1 and 2 of treatment (each cycle is 28 days)
  Defined as maximum observed plasma concentration
Pharmacokinetics (Tmax) for SY-4798 | Protocol-defined time points during Cycles 1 and 2 of treatment (each cycle is 28 days)
  Defined as time to maximum plasma concentration
Pharmacokinetics (AUC0-t) for SY-4798 | Protocol-defined time points during Cycles 1 and 2 of treatment (each cycle is 28 days)
  Defined as area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration
Pharmacokinetics (t½) for SY-4798 | Protocol-defined time points during Cycles 1 and 2 of treatment (each cycle is 28 days)
  Defined as the apparent plasma terminal phase disposition half-life
Pharmacokinetics (Cl/F) for SY-4798 | Protocol-defined time points during Cycles 1 and 2 of treatment (each cycle is 28 days)
  Defined as oral dose clearance

CONTACTS AND LOCATIONS:
Overall Officials: Yinghui Sun, PhD, Study Director — Shouyao Holdings (Beijing) Co. LTD
Locations (1):
- Shanghai East Hospital, Shanghai, China